CLINICAL TRIAL: NCT05037110
Title: Physical Activity and Sensory Trainings to Help COVID-19 Patients Recover From Persistent Smell and Taste Impairments - A Pilot Study
Brief Title: Physical Activity and Smell Trainings to Help Individuals With Coronavirus Disease (COVID-19) Recover From Persistent Smell and Taste Impairments - A Pilot Study
Acronym: CAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Ève Mathieu, Associate professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-374
Record Dates: First submitted 2021-09-02; First posted 2021-09-08 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: Olfactory training; Physical activity; Chemosensory impairments; Persistent smell impairment
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Exercise; Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity group (Experimental)
  Interventions: Behavioral: Physical activity
- Chemosensory training group (Experimental)
  Interventions: Other: Smell training
- Control group (No Intervention): For 12 weeks, continue the participant's routine (no intervention). This is done remotely. Then, every two weeks, complete an online follow-up questionnaire (15 minutes each).

INTERVENTIONS:
Behavioral: Physical activity — For 12 weeks, do 150 minutes of moderate physical activity per week and wear a smart watch to monitor this physical activity goal. This is done remotely. Then, every two weeks, attend a remote individual meeting with a kinesiologist using a secured application (15 minutes each). Each online meeting will contain the following steps: 1) Review of health and activities recorded by the activity watch/app provided to the participant; 2) Discussion on how to reach/maintain the physical activity goal in the coming weeks according to individual health status, facilitators and barriers; 3) Elaboration of the next 2-week action plan.
  Arms: Physical activity group
Other: Smell training — For 12 weeks, morning and evening, smell four odors namely eucalyptol, phenyl ethanol, citronellal, and eugenol, for a total of five minutes per session. For each smell training session, complete a short, online survey regarding the pleasantness and intensity of the smell. This is done remotely. Then, every two weeks, attend a remote individual meeting with a research professional using secured application (15 minutes each). Each online meeting will contain the following steps: 1) Review of smell training; 2) Discussion on how to reach/maintain the training protocol in the coming weeks according to individual health status, facilitators and barriers; 3) Elaboration of the next 2-week action plan.
  Arms: Chemosensory training group

SUMMARY:
The primary objective of this study is to identify efficient treatments to help those with chemosensory losses due to Coronavirus disease (COVID-19). To do so, 75 participants, men and women, aged 18 years old and above living in Canada will be recruited. Participants will be randomly assigned to one of the following three groups (25 in each group): physical activity, smell training, and control. Here is a quick summary of what participants in each group will have to do remotely during 12 weeks:

* Physical activity group: Engage in physical activity for 12 weeks and wear a smart watch daily. Attend a 15-minute virtual meeting with a research professional every two weeks, that is six times during the 12 weeks.
* Smell training group: Smell four odors twice a day for 12 weeks and evaluate their sensory perceptions via an online survey sent for each session specifically. Attend a 15-minute virtual meeting with a research professional every two weeks, that is six times during the 12 weeks.
* Control group: Not change their usual routine for 12 weeks. Complete an online 15-minute follow-up questionnaire every two weeks, that is six times over the 12 weeks.

In addition, within each group, 10 individuals from Montreal, Quebec will be randomly selected to complete additional assessments in the laboratory. To distinguish this subgroup, it is called the "in-person subgroup." Participants will be assessed at the beginning of the intervention period, immediately after the intervention period, and 12 weeks after the end of the intervention period. The assessments include various questionnaires on sociodemographic data, physical and mental health, lifestyle habits, sensory dysfunction, nutritional preferences, as well as self-administered smell and taste tests sent by mail. The in-person subgroup only will have to do the following additional assessments: smell and taste tests using special equipment (olfactometer, gustometer, electroencephalogram) and online questionnaires on food intake for the day.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old and above
* Have had COVID-19 diagnosed by laboratory tests
* Have recovered from COVID-19
* Have persistent problems with your sense of smell and/or taste due to COVID-19 in the past 3 months or more (priority to participants with only this complication)
* Have access to a computer and internet connection and be able to download the Zoom application
* Have access to a smart phone ("texting" and Bluetooth)
* Live in Canada

Exclusion Criteria:

* Do 150 minutes or more of physical activity that makes you out of breath every week
* Have limitations related to a training aiming at improving the sense of smell
* Have physical limitations that may limit physical activity
* Be part of another study that may influence the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in olfactory score on the 40-item University of Pennsylvania Smell Identification Test (UPSIT) at week 14 | Baseline and Week 14
  The UPSIT test is a validated self-administered test that assesses olfactory function. In this test, odorants are released when participants scratch the standardized odor-impregnated test booklet. After smelling the odor, participants identify the smell from a list of odorants. Possible scores range from 0 to 40, where a higher score means a higher olfactory function.
  Change = (Week 14 Score - Baseline Score)
Changes from Week 14 in olfactory score on the 40-item University of Pennsylvania Smell Identification Test (UPSIT) at Week 26. | Week 14 and Week 26
  The UPSIT test is a validated self-administered test that assesses olfactory function. In this test, odorants are released when participants scratch the standardized odor-impregnated test booklet. After smelling the odor, participants identify the smell from a list of odorants. Possible scores range from 0 to 40, where a higher score means a higher olfactory function.
  Change = (Week 26 Score - Week 14 Score)
Changes from Baseline in Gustatory Score on the 27-item Waterless Empirical Taste Test (WETT-SA) at Week 14 | Baseline and Week 14
  The WETT-SA test is a validated self-administered test that assesses gustatory function. Participants rub each strip, one at a time, on their tongues in a circular fashion. Then, they have to indicate what they tasted from a provided list of answers. Participants' answers are compared to an answer key and a higher score means a higher gustatory function
  Change = (Week 14 Score - Baseline Score)
Changes from Week 14 in Gustatory Score on the 27-item Waterless Empirical Taste Test (WETT-SA) at Week 26 | Week 14 and Week 26
  The WETT-SA test is a validated self-administered test that assesses gustatory function. Participants rub each strip, one at a time, on their tongues in a circular fashion. Then, they have to indicate what they tasted from a provided list of answers. Participants' answers are compared to an answer key and a higher score means a higher gustatory function
  Change = (Week 26 Score - Week 14 Score)
Changes from Baseline in Quality of Life on the 26-item World Health Organizations Quality of Life - Bref (WHOQoL-Bref) Questionnaire at Week 14 | Baseline and Week 14
  This is a validated questionnaire that assesses the quality of life. Each item is rated on a 5-point Likert scale. The higher the score, the higher the quality of life of the individual.
  Change = (Week 14 Results - Baseline Results)
Changes from Week 14 in Quality of Life on the 26-item World Health Organizations Quality of Life - Bref (WHOQoL-Bref) Questionnaire at Week 26 | Week 14 and Week 26
  This is a validated questionnaire that assesses the quality of life. Each item is rated on a 5-point Likert scale. The higher the score, the higher the quality of life of the individual.
  Change = (Week 26 Results - Week 14 Results)
Changes from Baseline in Food Preference on the Leeds Food Preference Questionnaire (LFPQ) at Week 14 | Baseline and Week 14
  LFPQ is a validated software that assesses food preferences. Participants are presented with food items. Participants have to indicate "How pleasant would it be to experience a mouthful of this food now?". Then, they are presented with two food items, and they have to decide which of those items they would prefer to eat now.
  This questionnaire is filled by participants in the in-person subgroup only.
  Change = (Week 14 Results - Baseline Results)
Changes from Week 14 in Food Preference on the Leeds Food Preference Questionnaire (LFPQ) at Week 26 | Week 14 and Week 26
  LFPQ is a validated software that assesses food preferences. Participants are presented with food items. Participants have to indicate "How pleasant would it be to experience a mouthful of this food now?". Then, they are presented with two food items, and they have to decide which of those items they would prefer to eat now.
  This questionnaire is filled by participants in the in-person subgroup only.
  Change = (Week 26 Results - Week 14 Results)
Changes from Baseline in Brain Responses Following Smell Stimulations at Week 14 | Baseline and Week 14
  Brain responses to smell stimulations an olfactometer will be recorded by an electroencephalogram.
  * The olfactometer is a device that gently blows different odors into the participant's nose at specific time intervals.
  * The electroencephalogram is a non-invasive device that records the electrical activity of the participant's brain. Electrical sensors are placed on helmet-like equipment that the participant wears while he/she smells or tastes samples.
  The brain activity is measured; smell event-related potentials (latency, duration, and amplitude) using an electroencephalogram are obtained.
  This procedure is done by participants in the in-person subgroup only.
  Change = (Baseline Results - Week 14 Results)
Changes from Baseline in Brain Responses Following Taste Stimulations at Week 14 | Baseline and Week 14
  Brain responses to taste stimulations using a gustometer will be recorded by an electroencephalogram.
  * The gustometer is a device that puts drops of different flavors on the participant's tongue at specific time intervals.
  * The electroencephalogram is a non-invasive device that records the electrical activity of the participant's brain. Electrical sensors are placed on helmet-like equipment that the participant wears while he/she smells or tastes samples.
  The brain activity is measured; taste event-related potentials (latency, duration, and amplitude) using an electroencephalogram are obtained.
  This procedure is done by participants in the in-person subgroup only.
  Change = (Baseline Results - Week 14 Results)
Changes from Week 14 in Brain Responses Following Smell Stimulations at Week 26 | Week 14 and Week 26
  Brain responses to smell stimulations using an olfactometer will be recorded by an electroencephalogram.
  * The olfactometer is a device that gently blows different odors into the participant's nose at specific time intervals.
  * The electroencephalogram is a non-invasive device that records the electrical activity of the participant's brain. Electrical sensors are placed on helmet-like equipment that the participant wears while he/she smells or tastes samples.
  The brain activity is measured; smell event-related potentials (latency, duration, and amplitude) using an electroencephalogram are obtained.
  This procedure is done by participants in the in-person subgroup only.
  Change = (Week 26 Results - Week 14 Results)
Changes from Week 14 in Brain Responses Following Taste Stimulations at Week 26 | Week 14 and Week 26
  Brain responses to taste stimulations using a gustometer will be recorded by an electroencephalogram.
  * The gustometer is a device that puts drops of different flavors on the participant's tongue at specific time intervals.
  * The electroencephalogram is a non-invasive device that records the electrical activity of the participant's brain. Electrical sensors are placed on helmet-like equipment that the participant wears while he/she smells or tastes samples.
  The brain activity is measured; taste event-related potentials (latency, duration, and amplitude) using an electroencephalogram are obtained.
  This procedure is done by participants in the in-person subgroup only.
  Change = (Week 26 Results - Week 14 Results)
Changes from Baseline in food intake on the four 24-hour dietary recall at Week 14 | Baseline and Week 14
  Validated web-based 24-hour dietary recalls assess the food intake of the participant over the past 24 hours. Participant reports what they have eaten over 24-hours, meal by meal. They are presented with different portion sizes from which they have to select the one corresponding to each food item. This will be completed on four different days within the week following the laboratory visit. Then, calories and macronutrients are calculated.
  These questionnaires are filled by participants in the in-person subgroup only.
  Change = (Week 14 Results - Baseline Results)
Changes from Week 14 in food intake on the four 24-hour dietary recall at Week 26 | Week 14 and Week 26
  Validated web-based 24-hour dietary recalls assess the food intake of the participant over the past 24 hours. Participant reports what they have eaten over 24-hours, meal by meal. They are presented with different portion sizes from which they have to select the one corresponding to each food item. This will be completed on four different days within the week following the laboratory visit. Then, calories and macronutrients are calculated.
  These questionnaires are filled by participants in the in-person subgroup only.
  Change = (Week 26 Results - Week 14 Results)

SECONDARY OUTCOMES:
Change from Baseline in physical activity level on the International Physical Activity Questionnaire (IPAQ) at week 14 | Baseline and Week 14
  IPAQ is a validated questionnaire. It assesses the physical activity level of participants over the past seven days. Based on the provided answer, a multiple of the estimated resting energy expenditure (METs) is calculated. Higher the METs value, the higher the physical activity level of the person.
  Change = (Week 14 Results - Baseline Results)
Change from Week 14 in physical activity level on the International Physical Activity Questionnaire (IPAQ) at week 26 | Week 14 and Week 26
  IPAQ is a validated questionnaire. It assesses the physical activity level of participants over the past seven days. Based on the provided answer, a multiple of the estimated resting energy expenditure (METs) is calculated. Higher the METs value, the higher the physical activity level of the person.
  Change = (Week 26 Results - Week 14 Results)

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The analyses will be centralized in Dr. Mathieu's laboratory and collaborations are welcomed.